CLINICAL TRIAL: NCT01917396
Title: Influence of Preoperative Enema Application on Return of Gastrointestinal Function After Elective Cesarean Section: A Randomized Controlled Study
Status: Approved for marketing | Type: Expanded Access
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, Obstetric and Gynecology, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Other Study IDs: Aşıcıoğlu 04
Record Dates: First submitted 2013-08-04; First posted 2013-08-06 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Bowel Sounds; Bowel Gass Passage
Keywords: caesarean, bowel, gass
MeSH Terms: interventions — sodium phosphate

INTERVENTIONS:
Drug: Fleet enema

SUMMARY:
The researchers investigate that use of preoperative enema to the effect postoperative bowel gas passage.

ELIGIBILITY:
Inclusion Criteria:

1. elective cesarean
2. no history of previous abdominal operation(except cs)

Exclusion Criteria:

1. Emergency cesarean delivery
2. Refusal to participate.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Egemen Ertaş, M.D., Principal Investigator — Tepecik Education and Research Hospital
Locations (1):
- Tepecik Education and Research Hospital,, Izmir, Yenisehir, Turkey (Türkiye)

REFERENCES:
- [Result] Lurie S, Baider C, Glickman H, Golan A, Sadan O. Are enemas given before cesarean section useful? A prospective randomized controlled study. Eur J Obstet Gynecol Reprod Biol. 2012 Jul;163(1):27-9. doi: 10.1016/j.ejogrb.2012.03.034. Epub 2012 Apr 17. PMID 22516178